CLINICAL TRIAL: NCT04433026
Title: B-natriuretic Peptide (BNP), Serum Troponin-I, and D-dimer as Risk Factors for In-hospital Death in Patients With COVID-19
Brief Title: BNP, Serum Troponin and D-dimer as Risk Factors in Patients With COVID-19
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Areej Osama Ali Mohammed Saleh, Resident physician, Assiut University
Other Study IDs: Cardiac markers in COVID-19
Record Dates: First submitted 2020-06-14; First posted 2020-06-16 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: N terminal pro B type natriuretic peptide (NTproBNP), D-Dimer, and serum Tropinin - I — Biomarkers detected in the serum of patients

SUMMARY:
To evaluate the role of N terminal pro B type natriuretic peptide (NTproBNP), D-Dimer, and Troponin - I as risk factors in COVID-19 patients and to correlate these markers with in-hospital death in patients with COVID-19

DETAILED DESCRIPTION:
Coronavirus disease-2019 (COVID-19), a contagious novel coronavirus now called severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2; formerly called 2019-nCoV).

Cardiac injury is a common condition among the hospitalized patients with COVID-19. It t was recently reported that 19.7% patients with COVID-19 had cardiac injury with more adverse clinical outcomes compared to those without cardiac injury (Shi S, et al, 2020) Fulminant myocarditis due to direct viral infection can certainly occur, but in patients with increased oxygen demands due to tachycardia and fever and reduced oxygen delivery due to hypotension and hypoxemia, COVID 19 disease can cause myocardial injury indirectly. Cytokines released during the acute infection can elicit activation of cells within pre-existing atherosclerotic lesions, augmenting thrombotic risk and risk of ischemic syndromes. Moreover, microvascular activation by cytokines can cause not only myocardial injury but can also harm other organ systems commonly involved in COVID-19 infections including the kidneys.(Peter,2020) Treatment in intensive care units (ICU) has become a major challenge; therefore, early recognition of severe forms is absolutely essential for timely triaging of patients. Several laboratory parameters may facilitate the assessment of disease severity. The recognized risk factors such as old age and underlying comorbidities-particularly cardiovascular diseases, diabetes, respiratory diseases, and other conditions (Zhou et al,2020) Several markers have been identified that modulate the course of COVID-19. The heart failure marker, N terminal pro B type natriuretic peptide (NT-proBNP), increased significantly during the course of hospitalization (Guo T, et al ,2020) The sensitivity of cardiac troponin testing that ensures it is one of the earliest and most precise indicators of end organ dysfunction. Cardiac troponin testing could prompt early initiation of measures to improve tissue oxygenation and perfusion.

COVID-19 infection is associated with intra-alveolar fibrin deposition, leading to lethal respiratory failure; reports suggesting that anticoagulation or fibrinolytic therapy can improve clinical outcomes (Wang J, et Al , 2020) ; case series implying that large percentages of severely affected COVID-19 patients suffer clinically significant thrombosis (Porfidia A , et al ,2020)

ELIGIBILITY:
Inclusion Criteria:

* patients with COVID-19 (moderate and severe cases) Different age groups

Exclusion Criteria:

* Patients who had stroke and acute myocardial infarction, malignant tumor, and pregnancy.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study initially enrolled 90 patients with COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of N-terminal pro-B type natriuretic peptide, troponin-I and D-dimer in COVID-19 patients | Baseline
  Measurement of the level of these markers in COVID-19 patients and collerate these measurements with early signs of cardiac injury in COVID-19 patients
Cardiac complications in COVID-19 patients associated with more adverse effects | Baseline
  Measurement of the level of N-terminal pro-B type natriuretic peptide, Troponin-I and D-dimer may help in detection of early signs of cardiac injury which in turn may help to minimize the risk of in-hospital deaths in COVID-19 patients

REFERENCES:
- [Background] Shi S, Qin M, Shen B, Cai Y, Liu T, Yang F, Gong W, Liu X, Liang J, Zhao Q, Huang H, Yang B, Huang C. Association of Cardiac Injury With Mortality in Hospitalized Patients With COVID-19 in Wuhan, China. JAMA Cardiol. 2020 Jul 1;5(7):802-810. doi: 10.1001/jamacardio.2020.0950. PMID 32211816
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Guo T, Fan Y, Chen M, Wu X, Zhang L, He T, Wang H, Wan J, Wang X, Lu Z. Cardiovascular Implications of Fatal Outcomes of Patients With Coronavirus Disease 2019 (COVID-19). JAMA Cardiol. 2020 Jul 1;5(7):811-818. doi: 10.1001/jamacardio.2020.1017. PMID 32219356
- [Background] Libby P. The Heart in COVID-19: Primary Target or Secondary Bystander? JACC Basic Transl Sci. 2020 Apr 10;5(5):537-542. doi: 10.1016/j.jacbts.2020.04.001. eCollection 2020 May. PMID 32292847
- [Background] Wang J, Hajizadeh N, Moore EE, McIntyre RC, Moore PK, Veress LA, Yaffe MB, Moore HB, Barrett CD. Tissue plasminogen activator (tPA) treatment for COVID-19 associated acute respiratory distress syndrome (ARDS): A case series. J Thromb Haemost. 2020 Jul;18(7):1752-1755. doi: 10.1111/jth.14828. Epub 2020 May 11. PMID 32267998
- [Background] Porfidia A, Pola R. Venous thromboembolism in COVID-19 patients. J Thromb Haemost. 2020 Jun;18(6):1516-1517. doi: 10.1111/jth.14842. No abstract available. PMID 32294289